CLINICAL TRIAL: NCT03567291
Title: An Open-Label, Long-Term Safety Study Including a Double-Blind, Placebo-Controlled, Randomized Withdrawal Period of TEV-50717 (Deutetrabenazine) for the Treatment of Tourette Syndrome in Children and Adolescents
Brief Title: Evaluation of Safety and Tolerability of Long-term TEV-50717 (Deutetrabenazine) for Treatment of Tourette Syndrome in Children and Adolescents
Acronym: ARTISTS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The parent trials did not meet the primary endpoints of reduction in motor and phonic tics.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Nuvelution TS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV50717-CNS-30047; 2016-000630-22 (EudraCT Number)
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tourette Syndrome
Keywords: adolescents; children
MeSH Terms: conditions — Tourette Syndrome | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TEV-50717- Part A (Experimental): All patients will undergo TEV-50717 dose titration in this study. Patients will receive 6 mg of TEV-50717 with food on the evening of day 1. The titration scheme and maximum dose will be determined by body weight and cytochrome P450 2D6 (CYP2D6) impairment status from the parent study.
  Interventions: Drug: TEV-50717
- TEV-50717- Part B RW (Experimental): TEV-50717 is administered during Part B Randomized Drug Withdrawal (RW) 2-week period.
  Interventions: Drug: TEV-50717
- Placebo- Part B RW (Placebo Comparator): Placebo is administered during Part B Randomized Drug Withdrawal (RW) 2-week period only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-50717 — 6, 9, and 12 mg oral tablets
  Other Names: deutetrabenazine, SD-809
  Arms: TEV-50717- Part A; TEV-50717- Part B RW
Drug: Placebo — Placebo comparator
  Arms: Placebo- Part B RW

SUMMARY:
This is an otherwise open-label, single-arm study that includes a 2-week, double-blind, placebo controlled, randomized drug withdrawal period followed by a 3 week blinded maintenance or re-titration, and then a maintenance period. This study aims to evaluate the safety and efficacy of TEV-50717 tablets in patients with tics associated with TS who have previously completed participation in any of the parent studies.

DETAILED DESCRIPTION:
This is an otherwise open-label, single-arm study (Part A) that includes a 2-week, double-blind, placebo controlled, randomized drug withdrawal period (Part B) followed by a 3 week blinded maintenance or re-titration (Part A resumed), and then a maintenance period. This study aims to evaluate the safety and efficacy of TEV-50717 tablets in patients with tics associated with TS who have previously completed participation in any of the parent studies (SD-809-C-17 [Phase 1b], TV50717-CNS 30046 [Phase 2/3], or TV50717-CNS 30060 [Phase 3]).

ELIGIBILITY:
Inclusion Criteria:

* Patient is younger than 18 years of age on day 1
* Patient weighs at least 44 pounds (20 kg)
* The patient's active tics are causing distress or impairment
* Patient is able to swallow study medication whole
* Patient is in good general health
* Women/girls of childbearing potential whose male partners are of childbearing potential must use contraception for the duration of the study -- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Patient is 18 years of age or older.
* Patient has a neurologic disorder other than TS that could obscure the evaluation of tics.
* The patient's predominant movement disorder is stereotypy (coordinated movements that repeat continually and identically) associated with autism spectrum disorder.
* Patient has a confirmed diagnosis of bipolar disorder, schizophrenia, or another psychotic disorder.
* Patient has clinically significant depression at screening or day 1. Note: Patients receiving antidepressant therapy may be enrolled if on a stable dose for at least 6 weeks before screening.
* Patient has a history of suicidal intent or related behaviors within 2 years of screening
* Patient has a history of a previous actual, interrupted, or aborted suicide attempt.
* Patient has a first-degree relative who has completed suicide.
* Patient has clinically significant obsessive-compulsive disorder (OCD) on day 1 that, in the opinion of the investigator, is the primary cause of impairment.
* Patient has received comprehensive behavioral intervention for tics for TS or cognitive behavioral therapy for OCD within 4 weeks of screening.
* Patient has received treatment with deep brain stimulation, transmagnetic stimulation, or transcranial direct current stimulation for reduction of tics within 4 weeks of the screening visit.
* Patient has an unstable or serious medical illness at screening or day 1
* Patients with a history of torsade de pointes, congenital long QT syndrome, bradyarrhythmias, or uncompensated heart failure.
* Patient has received a monoamine oxidase inhibitor within 14 days of the day 1 visit.
* Patient has participated in an investigational drug or device study (with the exception of Study SD-809-C-17, Study TV50717-CNS-30046, or Study TV50717-CNS-30060) and received IMP/intervention within 30 days or 5 drug half-lives of day 1, whichever is longer.
* The patient is a pregnant or lactating female, or plans to become pregnant during the study.
* Patient has a history of, or acknowledges, alcohol-related disorder in the previous 12 months -- Additional criteria apply, please contact the investigator for more information

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (76):
- United States (33):
  - Teva Investigational Site 046-0104, Dothan, Alabama
  - Teva Investigational Site 046-0107, Rogers, Arkansas
  - Teva Investigational Site 046-0126, Anaheim, California
  - Teva Investigational Site 046-0101, Sacramento, California
  - Teva Investigational Site 046-0111, San Diego, California
  - Teva Investigational Site 060-0160, Gainesville, Florida
  - Teva Investigational Site 060-0166, Gulf Breeze, Florida
  - Teva Investigational Site 060-0161, Miami, Florida
  - Teva Investigational Site 046-0115, Orlando, Florida
  - Teva Investigational Site 060-0153, Orlando, Florida
  - Teva Investigational Site 046-0114, St. Petersburg, Florida
  - Teva Investigational Site 046-0116, Atlanta, Georgia
  - Teva Investigational Site 060-0155, Chicago, Illinois
  - Teva Investigational Site 060-0164, Chicago, Illinois
  - Teva Investigational Site 046-0133, Naperville, Illinois
  - Teva Investigational Site 046-0128, Boston, Massachusetts
  - Teva Investigational Site 060-0170, Bridgeton, Missouri
  - Teva Investigational Site 046-0110, Saint Charles, Missouri
  - Teva Investigational Site 046-0134, Lincoln, Nebraska
  - Teva Investigational Site 046-0109, Voorhees Township, New Jersey
  - Teva Investigational Site 046-0124, New York, New York
  - Teva Investigational Site 060-0154, New York, New York
  - Teva Investigational Site 046-0102, Rochester, New York
  - Teva Investigational Site 046-0106, Oklahoma City, Oklahoma
  - Teva Investigational Site 060-0169, Charleston, South Carolina
  - Teva Investigational Site 060-0156, Nashville, Tennessee
  - Teva Investigational Site 046-0113, Dallas, Texas
  - Teva Investigational Site 060-0163, Fort Worth, Texas
  - Teva Investigational Site 046-0108, Houston, Texas
  - Teva Investigational Site 046-0120, San Antonio, Texas
  - Teva Investigational Site 046-0105, Orem, Utah
  - Teva Investigational Site 046-0118, Petersburg, Virginia
  - Teva Investigational Site 060-0162, Everett, Washington
- Argentina (4):
  - Teva Investigational Site 060-1407, Buenos Aires
  - Teva Investigational Site 060-1402, Buenos Aires
  - Teva Investigational Site 060-1403, La Plata
  - Teva Investigational Site 060-1404, Mendoza
- Teva Investigational Site 060-1802, Liverpool, Australia
- Canada (2):
  - Teva Investigational Site 046-0201, Ajax, Ontario
  - Teva Investigational Site 046-0202, Ottawa, Ontario
- Colombia (2):
  - Teva Investigational Site 060-1503, Bello
  - Teva Investigational Site 060-1504, Pereira
- Denmark (2):
  - Teva Investigational Site 046-0302, Herlev
  - Teva Investigational Site 046-0301, Odense
- Hungary (2):
  - Teva Investigational Site 060-0901, Budapest
  - Teva Investigational Site 060-0902, Szeged
- Italy (3):
  - Teva Investigational Site 060-1005, Cagliari
  - Teva Investigational Site 060-1001, Catania
  - Teva Investigational Site 060-1003, Naples
- Mexico (4):
  - Teva Investigational Site 060-1601, Culiacán
  - Teva Investigational Site 060-1603, León
  - Teva Investigational Site 060-1602, Monterrey
  - Teva Investigational Site 060-1604, Monterrey
- Poland (5):
  - Teva Investigational Site 060-1104, Gdansk
  - Teva Investigational Site 060-1101, Katowice
  - Teva Investigational Site 060-1105, Krakow
  - Teva Investigational Site 060-1102, Poznan
  - Teva Investigational Site 060-1103, Warsaw
- Russia (2):
  - Teva Investigational Site 046-0704, Tomsk
  - Teva Investigational Site 046-0703, Voronezh
- Serbia (3):
  - Teva Investigational Site 046-1702, Belgrade
  - Teva Investigational Site 046-1703, Belgrade
  - Teva Investigational Site 046-1701, Novi Sad
- South Korea (3):
  - Teva Investigational Site 060-1901, Seoul
  - Teva Investigational Site 060-1903, Seoul
  - Teva Investigational Site 060-1902, Seoul
- Spain (4):
  - Teva Investigational Site 046-0605, Madrid
  - Teva Investigational Site 046-0602, Madrid
  - Teva Investigational Site 046-0603, Málaga
  - Teva Investigational Site 046-0601, Seville
- Ukraine (6):
  - Teva Investigational Site 060-2003, Dnipropetrovsk
  - Teva Investigational Site 060-2001, Kharkiv
  - Teva Investigational Site 060-2002, Kharkiv
  - Teva Investigational Site 060-2007, Kiev
  - Teva Investigational Site 060-2005, Kyiv
  - Teva Investigational Site 060-2006, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 228 participants with Tourette Syndrome were enrolled after completing one of two eligible parent studies.
Pre-assignment Details: Period I (Part A) included a 28-week open-label period with a 7-week titration period followed by a maintenance period. Period II (Part B) included a two-week randomized drug withdrawal period (Weeks 28-30) in which participants were administered their current TEV50717 dose or placebo. Participants were re-titrated to TEV-50717 from Weeks 31-34. In Period III (Part A resumed), participants continued their open-label maintenance dose of TEV50717.
Groups:
- TEV-50717: All participants underwent TEV-50717 dose titration in this study. They received 6 mg of TEV-50717 with food on the evening of day 1. The titration scheme and maximum dose were determined by body weight and cytochrome P450 2D6 (CYP2D6) impairment status from the parent study.
- Randomized TEV-50717: Participants were randomized to their current dose of TEV-50717, which was administered during the Part B Randomized Drug Withdrawal (RW) 2-week period.
- Randomized Placebo: Participants were randomized to placebo, which was administered during the Part B Randomized Drug Withdrawal (RW) 2-week period only.
- TEV-50717 Re-titration and Maintenance: Participants who were randomized to placebo during the withdrawal period were re-titrated to their TEV-50717 maintenance dose. Participants who were randomized to TEV-50717 continued their maintenance dose.
Period: Period I
Arm/Group | TEV-50717 | Randomized TEV-50717 | Randomized Placebo | TEV-50717 Re-titration and Maintenance
Started | 228 | 0 | 0 | 0
Safety Set | 227 | 0 | 0 | 0
Intent to Treat Set | 228 | 0 | 0 | 0
Completed | 137 | 0 | 0 | 0
Not Completed | 91 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Terminated by sponsor | 44 | 0 | 0 | 0
Not completed — Missing or unknown | 7 | 0 | 0 | 0
Period: Period II
Arm/Group | TEV-50717 | Randomized TEV-50717 | Randomized Placebo | TEV-50717 Re-titration and Maintenance
Started | 0 | 91 | 46 | 0
Completed | 0 | 88 | 45 | 0
Not Completed | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Missing or unknown | 0 | 2 | 1 | 0
Period: Period III
Arm/Group | TEV-50717 | Randomized TEV-50717 | Randomized Placebo | TEV-50717 Re-titration and Maintenance
Started | 0 | 0 | 0 | 133
Completed | 0 | 0 | 0 | 48
Not Completed | 0 | 0 | 0 | 85
Not completed — Adverse Event | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Terminated by sponsor | 0 | 0 | 0 | 68
Not completed — Missing or unknown | 0 | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all enrolled participants.
Groups:
- All Participants: All participants underwent TEV-50717 dose titration in this study. They received 6 mg of TEV-50717 with food on the evening of day 1. The titration scheme and maximum dose were determined by body weight and cytochrome P450 2D6 (CYP2D6) impairment status from the parent study.
Arm/Group | All Participants
Number analyzed (Participants) | 228
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12 (2.59)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Participants: Male | 182
  Participants: Female | 45
  Participants: Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 186
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 197
  Black | 4
  Asian | 7
  Native American | 5
  Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (AEs) for Parts A & B Combined
Description: Adverse events were analyzed for all participants in Parts A & B combined as one group for this outcome measure. An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Incudes clinically significant changes such as changes in vital signs or lab values. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Day 1 to Week 55
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | TEV-50717
Number analyzed (Participants) | 227
Participants
  At least one adverse event | 161
  At least one serious adverse event | 2
  At least one severe adverse event | 6
  At least one AE related to investigational product | 95
  At least one adverse event leading to withdrawal | 14

2. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (AEs) in Part B (Period II)
Description: Adverse events were analyzed for Part B for this outcome measure. An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Incudes clinically significant changes such as changes in vital signs or lab values. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Weeks 28 to 30
Population: Population includes all participants who completed Period I, were randomized in Period II, and who were administered any study drug in the randomized withdrawal period, Part B (Period II).
Measure: Number; unit: Participants
Arm/Group | Randomized TEV-50717 | Randomized Placebo
Number analyzed (Participants) | 84 | 42
Participants
  At least one adverse event | 16 | 6
  At least one serious adverse event | 0 | 0
  At least one severe adverse event | 0 | 0
  At least one AE related to investigational product | 6 | 1
  At least one adverse event leading to withdrawal | 0 | 0

3. Primary Outcome: Change From Baseline in the Children's Depression Inventory Second Edition (CDI-2; Parent Version) Total Score
Description: Parents were asked to rate their child's behaviors in past 2 weeks on a 4-point Likert scale from "not at all" to "much or most of the time." It contains 2 subscales (emotional problems and functional problem). Total score: sum of 2 subscales, ranging from 0 to 51, with higher score indicating more depression-related behaviors.
Time Frame: Baseline, Weeks 2, 4, 8, 15, 28, 34, 41, 54, 55
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Units On A Scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 227
Units On A Scale
  CDI-2 Parent Version Week 2: number analyzed (Participants) | 221
  CDI-2 Parent Version Week 2 | -0.7 (4.26)
  CDI-2 Parent Version Week 4: number analyzed (Participants) | 221
  CDI-2 Parent Version Week 4 | -1.5 (4.39)
  CDI-2 Parent Version Week 8: number analyzed (Participants) | 217
  CDI-2 Parent Version Week 8 | -1.5 (5.0)
  CDI-2 Parent Version Week 15: number analyzed (Participants) | 210
  CDI-2 Parent Version Week 15 | -1.2 (5.79)
  CDI-2 Parent Version Week 28: number analyzed (Participants) | 145
  CDI-2 Parent Version Week 28 | -1.1 (5.52)
  CDI-2 Parent Version Week 34: number analyzed (Participants) | 118
  CDI-2 Parent Version Week 34 | -1.0 (6.08)
  CDI-2 Parent Version Week 41: number analyzed (Participants) | 95
  CDI-2 Parent Version Week 41 | -1.1 (5.92)
  CDI-2 Parent Version Week 54: number analyzed (Participants) | 48
  CDI-2 Parent Version Week 54 | -0.3 (5.83)
  CDI-2 Parent Version Week 55: number analyzed (Participants) | 47
  CDI-2 Parent Version Week 55 | -0.9 (4.34)

4. Primary Outcome: Change From Baseline in the Children's Depression Inventory Second Edition (CDI-2; Self-reported Version) Total Score
Description: CDI-2 self-report: 28-item questionnaire assessing depressive symptoms in children 7 to 17 years of age with basic reading and comprehension skills. Children were asked to choose 1 of 3 statements that most closely aligns with their feelings in past 2 weeks. It contains 6 subscales (emotional problem, negative mood/physical symptoms, negative self-esteem, functional problems, ineffectiveness, interpersonal problems). Total score: sum of all subscales scores, ranging from 0 to 56, with higher score indicating greater depression severity.CDI-2 parent: 17-item questionnaire administered to parents to assess depression-related behaviors observed in their children.
Time Frame: Baseline, Weeks 2, 4, 8, 15, 28, 34, 41, 54, 55
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units On A Scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 227
Units On A Scale
  CDI-2 Self-reported Version Week 2: number analyzed (Participants) | 198
  CDI-2 Self-reported Version Week 2 | -0.3 (3.41)
  CDI-2 Self-reported Version Week 4: number analyzed (Participants) | 203
  CDI-2 Self-reported Version Week 4 | -0.5 (3.57)
  CDI-2 Self-reported Version Week 8: number analyzed (Participants) | 205
  CDI-2 Self-reported Version Week 8 | -0.3 (4.35)
  CDI-2 Self-reported Version Week 15: number analyzed (Participants) | 204
  CDI-2 Self-reported Version Week 15 | -0.3 (4.83)
  CDI-2 Self-reported Version Week 28: number analyzed (Participants) | 142
  CDI-2 Self-reported Version Week 28 | 0.0 (4.65)
  CDI-2 Self-reported Version Week 34: number analyzed (Participants) | 117
  CDI-2 Self-reported Version Week 34 | -0.5 (4.61)
  CDI-2 Self-reported Version Week 41: number analyzed (Participants) | 94
  CDI-2 Self-reported Version Week 41 | -0.7 (4.74)
  CDI-2 Self-reported Version Week 54: number analyzed (Participants) | 48
  CDI-2 Self-reported Version Week 54 | -0.5 (4.01)
  CDI-2 Self-reported Version Week 55: number analyzed (Participants) | 47
  CDI-2 Self-reported Version Week 55 | -0.3 (4.52)

5. Primary Outcome: Change From Randomized Withdrawal Baseline (Week 28) in the Children's Depression Inventory Second Edition (CDI-2; Parent Version) Total Score at Week 30
Description: as for outcome 3
Time Frame: Week 28, Week 30
Population: Population includes all participants who completed Period I, were randomized in Period II, and who were administered any study drug in the randomized withdrawal period, Part B (Period II). Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Units On A Scale
Arm/Group | Randomized TEV-50717 | Randomized Placebo
Number analyzed (Participants) | 83 | 41
Units On A Scale | -0.2 (4.68) | 0.6 (3.62)

6. Primary Outcome: Change From Randomized Withdrawal Baseline (Week 28) in the Children's Depression Inventory Second Edition (CDI-2; Self-reported Version) Total Score at Week 30
Description: as for outcome 4
Time Frame: Week 28, Week 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units On A Scale
Arm/Group | Randomized TEV-50717 | Randomized Placebo
Number analyzed (Participants) | 82 | 39
Units On A Scale | -0.4 (3.30) | -0.6 (3.08)

7. Primary Outcome: Number of Participants Reporting Any Suicidal Ideation or Suicidal Behavior According to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS included responses for Suicidal Ideation or Suicidal Behavior in following 10 categories: 1 = Wish to be dead; 2 = Non-specific active suicidal thoughts; 3 = Active suicidal ideation with any methods (not plan) without intent to act; 4 = Active suicidal ideation with some intent to act, without specific plan; 5 = Active suicidal ideation with specific plan and intent; 6 = Preparatory acts or behavior; 7 = Aborted attempt; 8 = Interrupted attempt; 9 = Non-fatal suicide attempt; and 10 = Completed suicide. Number of participants with any suicidal ideation or suicidal behavior are reported. Any Suicidal ideation or Suicidal Behavior events reported as TEAEs along with all other reported TEAEs are included in the AE module.
Time Frame: Baseline, Weeks 2, 4, 8, 15, 28, 34, 41, 54, 55
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-50717
Number analyzed (Participants) | 227
Participants
  Baseline: number analyzed (Participants) | 225
  Baseline | 0
  Week 2: number analyzed (Participants) | 225
  Week 2 | 0
  Week 4: number analyzed (Participants) | 225
  Week 4 | 2
  Week 8: number analyzed (Participants) | 221
  Week 8 | 0
  Week 15: number analyzed (Participants) | 214
  Week 15 | 1
  Week 28: number analyzed (Participants) | 148
  Week 28 | 0
  Week 34: number analyzed (Participants) | 122
  Week 34 | 0
  Week 41: number analyzed (Participants) | 97
  Week 41 | 1
  Week 54: number analyzed (Participants) | 50
  Week 54 | 0
  Week 55: number analyzed (Participants) | 49
  Week 55 | 0

8. Primary Outcome: Number of Participants Reporting Any Suicidal Ideation or Suicidal Behavior According to the Columbia Suicide Severity Rating Scale (C-SSRS) at Randomized Withdrawal Baseline Visit (Week 28) and Week 30
Description: as for outcome 7
Time Frame: Week 28, Week 30
Population: Population includes all participants who completed Period I, were randomized in Period II, and who were administered any study drug in the randomized withdrawal period, Part B (Period II). Here, 'number analyzed' signifies participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized TEV-50717 | Randomized Placebo
Number analyzed (Participants) | 84 | 42
Participants
  Week 28: number analyzed (Participants) | 83 | 42
  Week 28 | 0 | 0
  Week 30: number analyzed (Participants) | 84 | 41
  Week 30 | 0 | 0

9. Secondary Outcome: Change From Baseline in the Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS)
Description: YGTSS rating scale is a semi-structured clinician rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic tics. YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 to severe). MTSS is the sum of the 5 items for motor tic severity and VTSS is the sum of the 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome. Baseline is defined as the last measurement on or prior to the first dose of the open-label study medication.
Time Frame: Baseline, Weeks 8, 15, 28, 41, 54, and 55
Population: ITT analysis set includes all participants enrolled in part I. Here, 'number analyzed' signifies participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 228
Units on a scale
  Week 8: number analyzed (Participants) | 217
  Week 8 | -6.9 (0.58)
  Week 15: number analyzed (Participants) | 211
  Week 15 | -7.8 (0.58)
  Week 28: number analyzed (Participants) | 145
  Week 28 | -6.2 (0.83)
  Week 41: number analyzed (Participants) | 92
  Week 41 | -8.3 (0.97)
  Week 54: number analyzed (Participants) | 47
  Week 54 | -6.5 (1.47)
  Week 55: number analyzed (Participants) | 45
  Week 55 | -4.3 (1.6)

10. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Clinical Global Impression (TS-CGI) Score
Description: The TS-CGI scale is a 7-point Likert scale that allows the clinician to use all available information to assess the impact of tics on the participant's quality of life. The TS-CGI is rated as follows: 1 (normal or no tics at all), 2 (borderline), 3 (mild), 4 (moderate), 5 (marked), 6 (severe), and 7 (extreme, incapacitating tics). Lower scores indicate better quality of life. Baseline is defined as the last measurement on or prior to the first dose of the open-label study medication.
Time Frame: Baseline, Weeks 8, 15, 28, 41, 54, and 55
Population: Data were not collected during Part B (Period II). ITT analysis set includes all participants enrolled in part I. Here, 'number analyzed' signifies participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 228
Units on a scale
  Week 8: number analyzed (Participants) | 216
  Week 8 | -0.7 (0.06)
  Week 15: number analyzed (Participants) | 209
  Week 15 | -0.7 (0.06)
  Week 28: number analyzed (Participants) | 144
  Week 28 | -0.6 (0.08)
  Week 41: number analyzed (Participants) | 91
  Week 41 | -0.6 (0.1)
  Week 54: number analyzed (Participants) | 47
  Week 54 | -0.8 (0.16)
  Week 55: number analyzed (Participants) | 47
  Week 55 | -0.4 (0.15)

11. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Patient Global Impression of Impact (TS-PGII) Score
Description: The TS-PGII is a single-item questionnaire that asks the participant to assess the degree of impact due to current tics (How much do your current tics disrupt things in your life?). The TS-PGII uses a 5-point scale, ranging from not at all (1) to very much (5), to assess overall response to therapy. Baseline is defined as the last measurement on or prior to the first dose of the open-label study medication.
Time Frame: Baseline, Weeks 8, 15, 28, 41, 54, and 55
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 228
Units on a scale
  Week 8: number analyzed (Participants) | 218
  Week 8 | -0.5 (0.07)
  Week 15: number analyzed (Participants) | 211
  Week 15 | -0.5 (0.08)
  Week 28: number analyzed (Participants) | 146
  Week 28 | -0.5 (0.09)
  Week 41: number analyzed (Participants) | 94
  Week 41 | -0.6 (0.12)
  Week 54: number analyzed (Participants) | 48
  Week 54 | -0.5 (0.16)
  Week 55: number analyzed (Participants) | 47
  Week 55 | -0.1 (0.14)

12. Secondary Outcome: Change From Baseline in the Child and Adolescent Gilles de la Tourette Syndrome - Quality of Life (C&A-GTS-QOL) Activities of Daily Living (ADL) Subscale Score
Description: C&A-GTS-QOL is a 27-item questionnaire that asks participant to assess the extent to which their quality of life is impacted by their symptoms. C&A-GTS-QOL contains 6 subscales (cognitive, coprophenomena, psychological, physical, obsessive-compulsive, and ADL) and uses a 5-point Likert scale ranging from no problem to extreme problem. Following 3 questions from 27-item questionnaire were assessed in ADL C&A-GTS-QOL subscale: Question 2 (Had difficulty with school or sport activities?), 24 (Felt you needed more help or support from other people?), and 26 (Had difficulty going out with other people?). Total score of ADL subscale ranged from 0 (no problem) to 12 (extreme problem). Lower score indicated better quality of life. Baseline is defined as the last measurement on or prior to the first dose of the open-label study medication.
Time Frame: Baseline, Weeks 6, 28, 34, 54
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 228
Units on a scale
  Week 6: number analyzed (Participants) | 203
  Week 6 | -4.9 (1.12)
  Week 28: number analyzed (Participants) | 135
  Week 28 | -4.4 (1.48)
  Week 34: number analyzed (Participants) | 106
  Week 34 | -5.9 (1.82)
  Week 54: number analyzed (Participants) | 44
  Week 54 | -2.7 (2.1)

13. Secondary Outcome: Change From Randomized Withdrawal Baseline (Week 28) in the Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) to Week 30
Description: YGTSS rating scale is a semi-structured clinician rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic tics. YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 to severe). MTSS is the sum of the 5 items for motor tic severity and VTSS is the sum of the 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome. The model is an ANCOVA model that includes fixed effects for treatment group. The randomized withdrawal baseline TTS and age group at baseline (2 levels: 6-11 years, 12-18 years) are included as covariates.
Time Frame: Week 28, Week 30
Population: All participants that completed Part 1, were randomized to Part 2, received at least one dose of study drug in the randomized withdrawal period and have an YGTSS TTS at both week 28 visit (randomized withdrawal baseline) and week 30 visit, and have a ≥25% reduction in the TTS from baseline in the parent study to week 28.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Randomized TEV-50717 | Randomized Placebo
Number analyzed (Participants) | 54 | 26
Units on a scale | 1.6 (0.86) | 2.0 (1.24)
Statistical Analysis 1: Comparison: Randomized TEV-50717 vs Randomized Placebo; Test type: Superiority; p = 0.78, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.4 to 2.6]

ADVERSE EVENTS:
Time Frame: Baseline to Week 55
Description: Adverse events were analyzed for participants in Parts A & B combined as one group per planned analysis. Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: All participants underwent TEV-50717 dose titration in this study. They received 6 mg of TEV-50717 with food on the evening of day 1. The titration scheme and maximum dose were determined by body weight and cytochrome P450 2D6 (CYP2D6) impairment status from the parent study.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/227
Serious Adverse Events (participants affected / at risk) | 2/227
Other Adverse Events (participants affected / at risk) | 108/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=227)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=227)
Vomiting (Gastrointestinal disorders) | 15 (30)
Pyrexia (General disorders) | 13 (13)
Nasopharyngitis (Infections and infestations) | 23 (33)
Weight increased (Investigations) | 22 (22)
Headache (Nervous system disorders) | 30 (55)
Somnolence (Nervous system disorders) | 28 (33)
Anxiety (Psychiatric disorders) | 17 (18)
Tic (Psychiatric disorders) | 15 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT03567291/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03567291/SAP_001.pdf